CLINICAL TRIAL: NCT04981613
Title: RCT Study on the Efficacy and Safety of a Novel Tripterygium Wilfordii Preparation in Reducing Proteinuria in Patients With Diabetic Nephropathy
Brief Title: Study on the Efficacy and Safety of a Novel Tripterygium Wilfordii Preparation in Reducing Proteinuria in Patients With Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYS2021-03-02-9
Record Dates: First submitted 2021-07-01; First posted 2021-07-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — kunxian

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Kunxian capsule (2# tid or 2# bid) + irbesartan tablet (150mg qd or 300mg qd) for 48 weeks
  Interventions: Drug: Kunxian capsule
- Control group (No Intervention): irbesartan tablet (150mg qd or 300mg qd) for 48 weeks

INTERVENTIONS:
Drug: Kunxian capsule — Kunxian capsule (2# tid or 2# bid) + irbesartan tablet (150mg qd or 300mg qd) for 48 weeks
  Arms: Experimental group

SUMMARY:
The investigators designed a randomized parallel controlled clinical study, selected 98 cases of diabetic nephropathy patients with urinary protein > 1g, randomly assigned into the Kunxian capsule + irbesartan group or irbesartan group, 48 weeks of treatment and follow-up, reduced levels of urinary protein and effective relief time, remission rate as the main end point, estimated glomerular filtration rate (eGFR) drop rate slope for secondary end points, safety events were also collected. To evaluate the efficacy and safety of Kunxian capsule combined with irbesartan in treatment of diabetic nephropathy compared with irbesartan alone.

ELIGIBILITY:
Inclusion Criteria:

* Conformed to the diagnostic criteria of diabetic nephropathy
* No gender limitation, age 18-85 years old, no fertility requirement temporarily
* eGFR: >30ml/min/1.73m2（CKD-EPI）
* Urine protein >1 g/day
* No glucocorticoids or/and immunosuppressive therapy was received within 3 months
* Patients volunteered to participate in this study and signed the informed consent

Exclusion Criteria:

* Combined with diabetic acute complications or acute kidney injury (AKI)
* Combined with other autoimmune diseases
* Primary and other secondary renal diseases
* Patients with hypotension (BP < 90/60mmHg) or bilateral renal artery stenosis who are not suitable for angiotensin receptor blockers (ARB) drugs
* There are contraindications to the use of kunxian capsules or allergic to any of the ingredients in kunxian capsules
* There are fertility requirements or pregnant, lactation patients
* Combined with malignant tumor, hepatitis, tuberculosis, HIV, serious infection, rheumatic disease, heart failure, chronic obstructive pulmonary disease (COPD) and other serious systemic diseases
* Kidney transplant or dialysis has been performed
* Clinicians deem it inappropriate, or patients are unwilling to sign informed consent, have poor compliance, have a history of mental illness, or cannot complete follow-up visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Changed levels of urinary protein, gram | 48 weeks
The effective remission time of urinary protein, day | 48 weeks
Urinary protein remission rate, % | 48 weeks

SECONDARY OUTCOMES:
24-hour urinary protein quantity, gram | 48 weeks
Urinary albumin/creatinine ratio | 48 weeks
eGFR decline rate slope | 48 weeks
Number of participants achieving end stage renal disease (ESRD) or requiring dialysis or kidney transplantation, or blood creatinine doubling, or renal death, or all-cause death, % | 48 weeks
Time of participants achieving end stage renal disease (ESRD) or requiring dialysis or kidney transplantation, or blood creatinine doubling, or renal death, or all-cause death, days | 48 weeks

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by bone marrow suppression, % | 48 weeks
Number of participants with treatment-related adverse events as assessed by liver damage, % | 48 weeks
Number of participants with treatment-related adverse events as assessed by infection, % | 48 weeks
Number of participants with treatment-related adverse events as assessed by gastrointestinal reactions, % | 48 weeks
Number of participants with treatment-related adverse events as assessed by skin damage, % | 48 weeks
Number of participants with treatment-related adverse events as assessed by reproductive toxicity (menorrhea or amenorrhea or infertility), % | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China